CLINICAL TRIAL: NCT03015012
Title: Using Personalized Nutrigenomics Testing to Mitigate Overweight/Obesity Risk in Two Distinct Patient Populations: A Multicentre Randomized Clinical Intervention Trial
Brief Title: Nutrigenomics, Overweight/Obesity and Weight Management Trial (NOW Trial)
Acronym: NOW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Collaborators: Nutrigenomix Inc. (Industry); East Elgin Family Health Team (Unknown); Canadian Transplant Association (Unknown)
Responsible Party: Principal Investigator, Janet Madill, Dr. Janet Madill, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 108511
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Transplant-Related Disorder; Overweight and Obesity
Keywords: Nutrigenomics; Genetics; Overweight; Obesity; Transplantation; Nutrition; Dietetics; BMI; Body Composition
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Nutrition Intervention (SNI) (Active Comparator): Transplant participants will receive standard nutrition counselling from a registered dietitian focused on strategies from the Canadian Diabetes Association's patient resource 'Just the Basics.' Nutrition counselling will focus on weight management. Individuals recruited from The East Elgin Family Health Team will complete the GLB Program. Transplant participants will receive a monthly follow-up email or phone call reviewing their nutrition and physical activity plan, until 12 months after baseline data collection. Reminders of lifestyle goals will be incorporated into the GLB Program for participants at the East Elgin Family Health Team.
  Interventions: Other: Standard Nutrition Intervention (SNI)
- Personalized Nutrigenomics Testing (PNT) (Experimental): Participants will receive nutrition counselling from a registered dietitian based on the results of their personalized nutrigenomics testing. Nutrition counselling will focus on weight management. Individuals recruited from The East Elgin Family Health Team will complete the GLB Program, but will be given personalized nutrition and physical activity advice based on the results of their nutrigenomics test. Transplant participants will receive a monthly follow-up email or phone call reviewing their nutrition and physical activity plan, until 12 months after baseline data collection. Reminders of lifestyle goals will be incorporated into the GLB Program for participants at the East Elgin Family Health Team.
  Interventions: Genetic: Personalized Nutrigenomics Testing (PNT)

INTERVENTIONS:
Genetic: Personalized Nutrigenomics Testing (PNT) — Participants will receive nutrition counselling from a registered dietitian based on the results of their personalized nutrigenomics testing. Nutrition and physical activity counselling will focus on weight management. Individuals recruited from The East Elgin Family Health Team will complete the GLB Program, but will be given personalized nutrition and physical activity advice based on the results of their nutrigenomics test. Transplant participants will receive a monthly follow-up email or phone call reviewing their nutrition and physical activity plan, until 12 months after baseline data collection. Reminders of lifestyle goals will be incorporated into the GLB Program for participants at the East Elgin Family Health Team.
  Arms: Personalized Nutrigenomics Testing (PNT)
Other: Standard Nutrition Intervention (SNI) — Transplant participants will receive standard nutrition counselling from a registered dietitian focused on strategies from the Canadian Diabetes Association's patient resource 'Just the Basics.' Nutrition and physical activity counselling will focus on weight management. Individuals recruited from The East Elgin Family Health Team will complete the standard GLB Program. Transplant participants will receive a monthly follow-up email or phone call reviewing their nutrition and physical activity plan, until 12 months after baseline data collection. Reminders of lifestyle goals will be incorporated into the GLB Program for participants at the East Elgin Family Health Team.
  Arms: Standard Nutrition Intervention (SNI)

SUMMARY:
The investigators hypothesize that compared to the provision of population-based lifestyle advice, providing DNA-based lifestyle advice via personalized nutrigenomics testing (PNT) to two distinct patient populations (Family Health Team patients receiving a lifestyle counselling intervention and transplant recipients) will lead to greater reductions in percent body fat. In addition, it will motivate them to adopt healthier dietary and physical activity habits through changes in attitudes and/or subjective norms and/or behavioural control, lead to greater fat loss (kg), increased percent lean mass and therefore improve health and quality of life outcomes for both patient populations. In addition, it is hypothesized that dietary strategies related to the intake of one or more dietary components of interest will mitigate post-transplant weight gain associated with three SNPs of interest.

This is a randomized clinical intervention trial involving a total of four groups of patients (n = 400). The two main patient groups include overweight or obese, stable transplant recipients and overweight or obese patients who are attending group counselling sessions at the East Elgin Family Health Team. Within these two main groups, there will be two sub-groups. Patients will be randomized to receive either PNT or standard nutrition intervention (SNI). Baseline data will be conducted consisting of a food frequency questionnaire and three-day food records using a validated multiple pass method. Bioelectrical Impedance Analysis (BIA) will be conducted to assess body composition and to derive percent body fat and lean mass. Weight and height will be measured using a weigh scale and stadiometer. Attitudes, subjective norms and behavioural control will be assessed using a Theory of Planned Behaviour Questionnaire. Those patients randomized to the PNT group will be instructed on a tailored nutrition care plan and physical activity recommendations based on their individual genetic profile. At the same time, the SNI group will be instructed on general nutrition and physical activity recommendations for weight loss, which include the use of dietary strategies from the standard tool ('Just the Basics') used by registered dietitians for transplant patients and the GLB program for patients attending the East Elgin Family Health Team sessions. Monthly email reminders or phone calls (depending on patient preference) will be sent to transplant recipients as a reminder of their nutrition and physical activity plan. Reminders of nutrition and physical activity goals for the Family Health Team participants are incorporated into the GLB program. Three months, six months and twelve months after baseline data collection and individual nutrition interventions, baseline data will be repeated. After the study is complete, participants in the SNI group will be offered a nutrigenomics report and consultation with a registered dietitian.

A paired t-test or repeated measures ANOVA will be used to assess within group change from baseline to each follow-up time point for: BMI, body fat, lean mass, and dietary intake. A repeated measures ANOVA will be used to test between group differences from baseline to each follow-up time point for: BMI, body fat, lean mass, and dietary intake. If significant mean differences are detected, a Tukey's post hoc test will be used to compare differences by group. Statistical significance will be determined by P < 0.05. General linear regression models will be used to assess interactions between each genotype of interest and each dietary component of interest on BMI and body composition from baseline to each follow-up time point.

DETAILED DESCRIPTION:
Hypotheses: Compared to the provision of population-based lifestyle advice, providing DNA-based lifestyle advice via personalized nutrigenomics testing (PNT) to two distinct patient populations (patients attending group counselling sessions at the East Elgin Family Health Team and transplant recipients) in which overweight and obesity are common concerns, will motivate them to adopt healthier dietary and physical activity habits via changes in attitudes and/or subjective norms and/or behavioural control, lead to greater fat loss, increased percent lean mass and therefore improve health and quality of life outcomes for both patient populations. It is also hypothesized that dietary strategies related to the intake of one or more dietary components of interest (protein, monounsaturated fat, polyunsaturated fat, total fat, sodium, carbohydrates, alcohol and calories) will mitigate post-transplant weight gain associated with the following SNPs: ACE (rs4343), FTO (rs1558902) and MC4R (rs571312).

Sample Size: No research to date has studied the aforementioned hypotheses. Previously published data assessing weight loss in a SNI group compared to a PNT group using a randomized clinical intervention model in a different population used a sample of n = 93 and an alpha < 0.05 to find statistical significance after 3-7 month follow-up. Similarly, nutrigenomics research in the ACE gene (rs4343) found statistical significance using a sample of n = 104 and an alpha < 0.05. A sample size calculation with 80% power and an alpha of 0.05 indicated that 37 participants per group (n = 148 total) are needed to detect significant differences between groups for changes in body fat percentage (primary outcome). Since it is feasible for this research, a larger sample size goal (n = 400) will be used to increase power and draw meaningful inferences from the data. There will be 100 participants in each patient group (n = 200 in SNI group, n = 200 in PNT group) in this landmark study.

Design and Methods: Participants will be recruited from the Canadian Transplant Association (CTA) meetings with the assistance of the Director, Sandra Holdsworth (transplant recipients; n = 200) and from the Group Lifestyle Balance Program (GLB Program) through the East Elgin Family Health Team (GLB; n = 200) for this randomized clinical intervention trial. Word-of-mouth recruitment is also expected. This trial involves a total of four groups of patients. The two main patient groups include overweight or obese (BMI ≥ 25 kg/m^2), stable transplant recipients greater than or equal to one year post-transplant, and overweight or obese (BMI ≥ 25 kg/m^2) patients who are attending the GLB program at the East Elgin Family Health Team. Within these two main patient groups, there will be two sub-groups (n = 100 per sub-group). Patients will be randomized to receive either PNT or standard nutrition intervention (SNI) based on strategies from the standard teaching tool used by dietitians in both patient populations: 'Just the Basics' - developed by the Canadian Diabetes Association for transplant participants. Participants from the East Elgin Family Health Team, will participate in the GLB Program and will either complete the standard program (SNI Group) + receive population-based nutrition and physical activity recommendations or will complete a modified GLB program + receive personalized nutrition and physical activity recommendations based on their genetics (PNT Group). Baseline data will be conducted consisting of a food frequency questionnaire and three-day food records using a validated multiple pass method. Bioelectrical Impedance Analysis (BIA) will be conducted to assess body composition and to derive percent and kg body fat and lean mass. Weight and height will be measured using a weigh scale and stadiometer. Surveys will be completed by participants to assess several demographic characteristics, as well as key components of the Theory of Planned Behaviour. Those patients randomized to the PNT group will be instructed on a tailored nutrition care plan and physical activity goal based on their individual genetic profile. At the same time, the SNI group will be instructed on general nutrition and physical activity recommendations for weight loss. A survey based on the Theory of Planned Behaviour will be administered before and after participants receive their nutrition and physical activity advice. These components are needed so that we can assess whether or not social and built environment factors, subjective norms, attitudes and behavioural control influence change in dietary intake. Monthly email or phone call reminders (depending on participant preference) will be sent to participants as a reminder of their nutrition and physical activity plan for transplant recipients. For East Elgin Family Health Team participants, reminders of the nutrition and physical activity plan will be incorporated into the GLB Program. Three months, six months and twelve months after baseline data collection and individual nutrition interventions, baseline data will be repeated. After the study is complete, participants in the SNI group will be offered a nutrigenomics test and consultation with a registered dietitian.

Statistical Analysis: A paired t-test or repeated measures ANOVA will be used to assess within group change from baseline to each of the follow-up time points for: BMI, body fat, lean mass, water weight, TPB components, dietary intake (protein, total fat, saturated fat, unsaturated fat, carbohydrates, alcohol, calories and sodium), and physical activity. A repeated measures ANOVA will be used to test between group differences from baseline to each of the follow-up time points for: BMI, body fat, lean mass, water weight, TPB components, dietary intake (protein, total fat, saturated fat, unsaturated fat, carbohydrates, alcohol, calories and sodium) and physical activity. If significant mean differences are detected, a Tukey's post hoc test will be used to compare differences by group. Statistical significance will be determined by P < 0.05. General linear regression models will be used to assess the effect of each genotype of interest (ACE rs4343, MC4R rs573112, FTO rs1558902) and the impact of each dietary component of interest (protein, total fat, saturated fat, unsaturated fat, carbohydrates, alcohol, calories and sodium) on BMI and body composition from baseline to each follow-up time point. We will control for age, sex, ethnicity, immunosuppressive medications (transplant recipients) and baseline body composition and BMI. IBM SPSS Statistics, version 21.0 will be used for the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* TRANSPLANT PATIENTS: Adults greater than or equal to age 18, non-pregnant, non-lactating, attending Canadian Transplant Association meetings, BMI ≥ 25kg/m2, ≥1 year stable (not being treated for transplant rejection or infection) post-transplant, having access to a computer with email or a telephone at least one day per week and English speaking.
* LIFESTYLE INTERVENTION PROGRAM (GLB) PATIENTS: Adults greater than or equal to age 18, non-pregnant, non-lactating, BMI ≥ 25kg/m2, having access to a computer with email or a telephone at least one day per week and English speaking.

Exclusion Criteria:

* TRANSPLANT PATIENTS: Patients with BMI <25 kg/m2, unwilling to undergo PNT, unable to provide consent, undergoing treatment for transplant rejection or infection, not English speaking, without access to a computer with email or a telephone at least one day per week and/or <1 year post-transplant, seeing another healthcare provider for weight loss advice outside of this study
* LIFESTYLE INTERVENTION PROGRAM (GLB) PATIENTS: Patients with BMI <25 kg/m2, unwilling to undergo PNT, unable to provide consent, not English speaking, without access to a computer with email or a telephone at least one day per week, seeing another healthcare provider for weight loss advice outside of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in Body Fat Percentage | 3 months, 6 months, 12 months
  Change in body composition (body fat percentage as the primary outcome) will be assessed using BIA which will provide information on fat mass, lean mass, and water weight

SECONDARY OUTCOMES:
Change in Dietary Intake | 3 months, 6 months, 12 months
  Change in dietary intake will be assessed using pre- and post- dietary data collected using 3-day food records, and a past-month online food frequency questionnaire.
Change in Physical Activity | 3 months, 6 months, 12 months
  Change in physical activity will be assessed using pre- and post- physical activity data collected using a 7-day physical activity recall. Metabolic equivalents will then be calculated from this data.
Change in Attitudes, Subjective Norms and Behavioural Control | Pre- and post- lifestyle intervention (baseline), 3 months, 6 months, 12 months
  Change in these key components of the Theory of Planned Behaviour (TPB) will be assessed using a TPB questionnaire.
Change in Body Composition | 3 months, 6 months, 12 months
  Change in body composition will be assessed using BIA which will provide information on fat mass, lean mass, and water weight
BMI | 3 months, 6 months, 12 months
  Change in BMI will be measured using weight and height data collected using a weigh scale and stadiometer
Weight | 3 months, 6 months, 12 months
  Change in weight will be measured using a weigh scale

OTHER OUTCOMES:
Nutrigenomics Interactions | 3 months, 6 months, 12 months
  Nutrigenomics (nutrition-genetic) interactions between ACE gene variants at rs4343, FTO gene variants at rs1558902 (in strong linkage disequilibrium with rs9939609) and MC4R (rs571312) to mitigate risk of post-transplant weight gain will be assessed for transplant recipients in the PNT group.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Madill, PhD, Principal Investigator — Brescia University College at Western University
Locations (2):
- Canada (2):
  - East Elgin Family Health Team, Aylmer, Ontario
  - Brescia University College, London, Ontario

IPD SHARING:
Plan to Share IPD: No
IPD will only be available to the current research team.

REFERENCES:
- [Background] Horne J, Gilliland J, O'Connor C, Seabrook J, Hannaberg P, Madill J. Study protocol of a pragmatic randomized controlled trial incorporated into the Group Lifestyle Balance program: the nutrigenomics, overweight/obesity and weight management trial (the NOW trial). BMC Public Health. 2019 Mar 15;19(1):310. doi: 10.1186/s12889-019-6621-8. PMID 30876469
- [Derived] Horne JR, Gilliland JA, Vohl MC, Madill J. Exploring Attitudes, Subjective Norms and Perceived Behavioural Control in a Genetic-Based and a Population-Based Weight Management Intervention: A One-Year Randomized Controlled Trial. Nutrients. 2020 Dec 8;12(12):3768. doi: 10.3390/nu12123768. PMID 33302460
- [Derived] Horne J, Gilliland J, O'Connor C, Seabrook J, Madill J. Enhanced long-term dietary change and adherence in a nutrigenomics-guided lifestyle intervention compared to a population-based (GLB/DPP) lifestyle intervention for weight management: results from the NOW randomised controlled trial. BMJ Nutr Prev Health. 2020 May 21;3(1):49-59. doi: 10.1136/bmjnph-2020-000073. eCollection 2020. PMID 33235971
- [Derived] Horne JR, Gilliland J, Leckie T, O'Connor C, Seabrook JA, Madill J. Can a Lifestyle Genomics Intervention Motivate Patients to Engage in Greater Physical Activity than a Population-Based Intervention? Results from the NOW Randomized Controlled Trial. Lifestyle Genom. 2020;13(6):180-186. doi: 10.1159/000510216. Epub 2020 Oct 1. PMID 33002888
- [Derived] Horne JR, Gilliland JA, O'Connor CP, Seabrook JA, Madill J. Change in Weight, BMI, and Body Composition in a Population-Based Intervention Versus Genetic-Based Intervention: The NOW Trial. Obesity (Silver Spring). 2020 Aug;28(8):1419-1427. doi: 10.1002/oby.22880. PMID 32935529